CLINICAL TRIAL: NCT07150065
Title: Efficacy of Levofloxacin Versus Ciprofloxacin in the Treatment of Childhood Typhoid Fever
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avicenna Medical College Lahore (Other)
Responsible Party: Principal Investigator, Muhammad Iqbal, Principal Investigator, Avicenna Medical College Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 107
Record Dates: First submitted 2025-08-17; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Typhoid; Fever
Keywords: ciprofloxacin; children; enteric fever; levofloxacin
MeSH Terms: conditions — Typhoid Fever; Fever | interventions — Levofloxacin; Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A with oral 200 mg levofloxacin tablet (Active Comparator): Group A included 180 participants. They were given oral 200 mg levofloxacin tablet. All children were followed-up pediatric wards for 7 days. If fever was resolved within 5 days (body temperature falls <99oF and remain stable for at least 5 days), then efficacy was labeled. Total time required to resolve fever i.e. body temperature <99oF in all children was also noted.
  Interventions: Drug: Levofloxacin
- Group B with oral 900-1,000 mg ciprofloxacin tablet (Active Comparator): . In group B, children were given oral 900-1,000 mg ciprofloxacin tablet. All children were followed-up pediatric wards for 7 days. If fever was resolved within 5 days (body temperature falls <99oF and remain stable for at least 5 days), then efficacy was labeled. Total time required to resolve fever i.e. body temperature <99oF in all children was also noted
  Interventions: Drug: ciprofloxacin

INTERVENTIONS:
Drug: Levofloxacin — Oral 200 mg levofloxacin tablet
  Arms: Group A with oral 200 mg levofloxacin tablet
Drug: ciprofloxacin — Oral 900-1,000 mg ciprofloxacin tablet
  Arms: Group B with oral 900-1,000 mg ciprofloxacin tablet

SUMMARY:
Sample size of 360 children with typhoid fever were enrolled and randomly divided in two groups. All the children were enrolled in the trial from Pediatrics emergency. Informed consent was obtained from parents. Demographics (name, age of child, sex of the child, duration of fever, weight, season, socioeconomic status and residence) were noted. Then children were admitted and randomly divided in two groups by using lottery method. In group A, children were given oral 200 mg levofloxacin tablet. In group B, children were given oral 900-1,000 mg ciprofloxacin tablet. All children were followed-up pediatric wards for 7 days. If fever was resolved within 5 days (body temperature falls <99oF and remain stable for at least 5 days), then efficacy was labeled. Total time required to resolve fever i.e. body temperature <99oF in all children was also noted. All this information was recorded

ELIGIBILITY:
Inclusion Criteria:

* Children of age 1-12 years
* Typhoid fever
* Confirmed on blood culture

Exclusion Criteria:

* Recurrent typhoid within 3 months
* Intestinal perforation
* Evidence of progressive or complicated disease
* Inability to swallow oral medication
* Hypersensitivity to trial drugs
* Already taken fluoroquinolone, third generation cephalosporin or macrolide in last week

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2025-02-07 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
Total time required to resolve fever | 5 days
  Clinical efficacy involved resolution of fever within 5 days (body temperature falls <99oF and remain stable for at least 5 days). Total time required to resolve fever i.e. body temperature <99oF in all children was also noted.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Aneela Zareen, MBBS FCPS, Study Director — Avicenna Medical And Dental College
Locations (1):
- Avicenna Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No